CLINICAL TRIAL: NCT04892485
Title: Relationship of Skeletal Muscle Thickness, Strength, and Diaphragm Function in Adults With CF
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Berrin Ceyhan, Professor, Marmara University
Other Study IDs: 09.2016.341
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Cystic Fibrosis
Keywords: CF, nutritional status, peripheral muscle thickness, peripheral muscle strength, diaphragm thickening fraction
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- CF patients
- Controls

SUMMARY:
31 CF patients and 23 healthy sex and age-matched volunteers were enrolled. All subjects underwent pulmonary function tests, 6-minute walking tests. Body Mass Index and Fat Free Mass Index were measured via a body composition analyser. Diaphragm ultrasonography (to measure thickening fraction), quadriceps femoris muscle ultrasonography were performed. A dynamometer was used to measure each subjects handgrip strength.

ELIGIBILITY:
Inclusion Criteria:

* CF diagnosed
* Age 18 and above

Exclusion Criteria:

* Having a pulmonary flare up within the previous month
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult CF patients and healty age sex matched controls
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Muscle Thickness, Strength and Diaphragm Thickening Fraction of CF Patients | 2 months
  Measured via USG and handheld dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Berrin Ceyhan, Prof, Study Chair — Marmara University
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided